CLINICAL TRIAL: NCT03590249
Title: Effects of a Single Osteopathic Manipulative Treatment (OMT) on Intraocular Pressure (IOP) Reduction
Acronym: OMT/IOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hollis King, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160684
Record Dates: First submitted 2018-07-04; First posted 2018-07-18 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Glaucoma
Keywords: osteopathic manipulative treatment
MeSH Terms: conditions — Glaucoma | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: The design of this preliminary pilot trial is a double-masked (blind), randomized, No Treatment-controlled, parallel group design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The practitioner providing the OMT or No Treatment will not be involved in collecting data for each subject. The practitioner(s) and technicians collecting the data will not be involved in any aspect of the procedure performed (OMT or No Treatment) on the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulative Treatment (OMT) (Experimental): Osteopathic manipulation involves a number of different manual (hands-on) techniques. These include muscle inhibition (applying pressure to a muscle to induce relaxation); myofascial release (applying pressure to the fascia and moving it toward/away from a strain); muscle energy stretch (contraction of a stretching muscle); counterstrain (shortening a strained muscle); facilitated positional release (moving a vertebra into a restriction and applying a gentle compression); osteopathy in the cranial field (balancing the cranial tissue); balanced ligamentous tension/ligamentous articular strain (moving a joint into ease to release tension in the ligament); one or all of these techniques may be used. Participants will be positioned on an exam table supine, seated, lateral decubitus, prone, or in their position of greatest comfort for the procedure.
  Interventions: Procedure: Osteopathic Manipulative Treatment
- No Intervention (No Intervention): Participants in the No Intervention arm will undergo the planned assessments, but not receive any intervention.

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Osteopathic manipulation involves a number of different manual (hands-on) techniques. These include muscle inhibition (applying pressure to a muscle to induce relaxation); myofascial release (applying pressure to the fascia and moving it toward/away from a strain); muscle energy stretch (contraction of a stretching muscle); counterstrain (shortening a strained muscle); facilitated positional release (moving a vertebra into a restriction and applying a gentle compression); osteopathy in the cranial field (balancing the cranial tissue); balanced ligamentous tension/ligamentous articular strain (moving a joint into ease to release tension in the ligament); one or all of these techniques may be used. Participants will be positioned on an exam table supine, seated, lateral decubitus, prone, or in their position of greatest comfort for the procedure. Treatment will last approximately 45 minutes.
  Arms: Osteopathic Manipulative Treatment (OMT)

SUMMARY:
Glaucoma is a group of eye diseases, which in most cases produce increased pressure within the eye (intraocular pressure or IOP). Over time, the elevated IOP causes damage to the optic nerve, which can then lead to visual loss and if unchecked, to complete blindness over the course of years. OMT has been shown to affect cranial structure physiology including the possibility of lowering IOP by improving the drainage of intraocular fluid. This randomized study is designed to obtain data to evaluate the effect of OMT on IOP lowering and, if supportive, provide preliminary data for larger clinical trials.

DETAILED DESCRIPTION:
The design of this preliminary pilot trial to be conducted is a double-masked (blind), randomized, No Treatment-controlled, parallel group design to determine the IOP-lowering efficacy and safety of a single osteopathic manipulative treatment (OMT) on intraocular pressure (IOP) in un-medicated confirmed ocular hypertensive (OHT), glaucoma suspect, or subjects who have been diagnosed with glaucoma but who have gone through a medically supervised medication washout period or 4 weeks.

Potential subjects responding to recruitment who are currently on IOP lowering medication will be prescreened and if interested in proceeding will undergo a 4 week medication washout period. Potential subjects not on IOP lowering medication will proceed directly to the Baseline screening visit.

All subjects will be seen for a Baseline Screening Visit followed by a second Baseline Enrollment Visit, during which subjects must satisfy all inclusion criteria and their IOP must qualify in at least one (1) eye, the same eye, at all time points. Qualified subjects will be scheduled for a Study Day 3 Visit. Subjects whose IOP still qualifies at the Visit 3 time point will be randomized in a 1:1 ratio to receive OMT or No Treatment followed by IOP measurements and +7.5 HR (4 PM [± 1 hour]) post-OMT or No Treatment. Follow-up visits will be conducted at Visit 4 (1 day following OMT vs No Treatment), and Visit 5 (1 week following OMT vs No Treatment). Both Visit 4 and Visit 5 will have IOP measured twice.

ELIGIBILITY:
Subject inclusion criteria:

1. Subjects will be of either sex, age 18 years or older, and of any race or eye color.
2. Subjects with confirmed ocular hypertension (OHT), glaucoma suspects or diagnosed with primary open-angle glaucoma whose IOP was ≥ 20 mmHg at two measurements separated by at least 3 months. If subject already on IOP lowering medication and goes through the 4 week washout, they must still have initial IOP ≥ 20 mmHg at the Baseline I screening visit.
3. Subjects who do not have visual field defect(s), as determined by Visual Field Analysis within the last year such as "blind spots" and other visual image distortions from normal vision.
4. Subjects who do not have abnormal cupping of the optic nerve head.
5. Subjects who do not have narrow angles as determined by gonioscopy (must be at least angle grade 2 to 3; Shaffer Classification Scale) recorded in the subject's patient record or as determined by biomicroscopy.
6. Subjects who have not been treated with ocular hypotensive agents (or, if they have been treated, not for at least the preceding 4 weeks before Baseline I Screening).
7. Subjects must satisfy all informed consent requirements.
8. Subjects whose mean IOP measurements in at least one (1) eye, the same eye(s), must be:

   * Greater than or equal to 20 mmHg at the 8:00 AM time-point on the Screening and Enrollment Visits (1 and 2) and
   * Greater than or equal to 19 mmHg at the 5 PM time-points on the Screening and Enrollment Visits (1 and 2).

Subject exclusion criteria:

1. Subjects who have had any traumatic brain injury or head trauma, which resulted in upper-spinal fusion which requires metal or plastic screws or plates and/or cranial bone surgery, which involves penetration of the cranial bones and/or implantation of a metal plate.
2. Subjects who have a concurrent diagnosis of cancer or metastatic disease affecting the head and neck.
3. Subjects who are less than 18 years old.
4. Subjects who are lactating, pregnant, or plan to become pregnant in the time planned for the study, to be confirmed by a urine pregnancy if the woman is still menstruating.
5. Subjects who have a history of chronic or recurrent severe inflammatory eye disease (e.g., scleritis - inflammation of the white part of the eye or uveitis - eye redness, pain and blurred vision) in either eye as determined by patient history and/or examination.
6. Subjects who have a history of clinically significant or progressive retinal disease in either eye such as retinal degeneration (which is the breakdown of the light-sensitive cells in retina), diabetic retinopathy (involves changes to retinal blood vessels that can cause them to bleed or leak fluid), or retinal detachment which is separation of the retina from the layer of cells behind it with permanent field loss as determined by patient history and/or examination.
7. Subjects who have a history of serious ocular trauma in either eye within the past six (6) months as determined by patient history and/or examination.
8. Subjects who have had intraocular surgery in either eye within the past six (6) months as determined by patient history and/or examination.
9. Subjects who have had ocular laser surgery, which is the use of a laser beam to make a very small hole in the eye tissue (also known as Lasik) in either eye within the past three (3) months as determined by patient history and/or examination.
10. Subjects who have a history of ocular infection or ocular inflammation in either eye within the past three (3) months as determined by patient history and/or examination.
11. Subjects who have any abnormality preventing reliable applanation tonometry of either eye (e.g., keratoconus (a thinning of the cornea), cornea (eyes outer most layer) or conjunctiva (the mucous membrane that covers the front of the eye and lines the inside of the eyelids) scarring.
12. Subjects who have less than a thirty (30) days stable dosing regimen before the Screening and Enrollment Visits (Visits 1 and 2) of any non-ocular medications that may affect IOP, administered by any route and used on a chronic basis. These may include, but are not limited to, alpha agonists, beta-blockers, calcium channel blockers, antimuscarinic agents, and phenothiazines.
13. Subjects who have other treatments and/or surgeries unrelated to the eye condition scheduled in the time planned for the study.
14. Subjects who are allergic to Latex, PABA, Proparacaine, or Fluorescein.
15. Subjects who have had prior surgical or laser treatment for the purpose of lowering their IOP.
16. Subjects who currently have systemic infections resulting in fever or immunosuppression.
17. Subjects who have had previous manual medicine or manual therapy with manually guided gentle forces to realign musculoskeletal imbalances or relax strained muscles such as osteopathic manipulative treatment (OMT), chiropractic manipulation, massage within the last 2 months.
18. Subjects who are unable to give appropriate informed consent due to mental or other limitations.
19. Additionally, the Principal Investigator may declare any subject ineligible for a valid medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure Change | 1-day and 1-week post-intervention or no intervention
  All vision data are collected by Hamilton Glaucoma Center trained research staff and physicians. The primary outcome measure, IOP (Goldman tonometry) will be collected and read by two people in the "masked IOP" procedure and the readings will be averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Hollis H King, DO, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Shiley Eye Center, University of California, San Diego, La Jolla, California, United States